CLINICAL TRIAL: NCT05548608
Title: Effect of Different Injury Mechanism on Lumbar Proprioception in Patients With Lumbar Spinal Stenosis: an Observational Healthy Controlled Study
Brief Title: Lumbar Proprioception in Patients With Lumbar Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Şule ŞİMŞEK, PhD faculty member, Pamukkale University
Other Study IDs: 28.07.2020/14
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Lumbar spinal stenosis; proprioception; reposition error
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (Healthy control): Group I consists of patient relatives and patients who applied to the outpatient clinic for another ailment.
  Interventions: Other: Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively.
- Group II (chronic low back pain due to LSS ): Group II consisted of patients diagnosed with LSS and confirmed by MRI findings.
  Interventions: Other: Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively.
- Group III (undergoing surgery due to LSS ): Participants who had surgery for LSS at least 3 months ago were included in Group III.
  Interventions: Other: Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively.

INTERVENTIONS:
Other: Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively. — Target positions of reposition error were: 30º forward bending and 15º backward bending in sitting and standing.

SUMMARY:
The primary aim of this study was to compare spinal proprioception in patients with Lumbal Spinal Stenosis (LSS) (with or without surgery) and healthy controls. A secondary aim was to investigate the effect of pain at target positions where repositioning error (RE) was assessed and TLF flexibility on spinal proprioception deficiency.This cross-sectional and healthy controlled study was conducted in patients with LSS. Participants will be grouped as: Healthy control (Group I), chronic low back pain due to LSS (Group II) and undergoing surgery due to LSS (Group III). Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively. Target positions of reposition error were: 30º forward bending and 15º backward bending in sitting and standing.

DETAILED DESCRIPTION:
This cross-sectional and healthy controlled study was conducted in patients with LSS. Participants will be grouped as: Healthy control (Group I), chronic low back pain due to LSS (Group II) and undergoing surgery due to LSS (Group III). Reposition error (RE), pain at target positions of RE and flexibility of the TLF were assesed with iphone tiltmeter app, VAS and goniometric platform, respectively. Target positions of reposition error were: 30º forward bending and 15º backward bending in sitting and standing.

The general study inclusion criteria were as follows: age between 20 and 50 years and not having had lower extremity surgery.

In addition to the general inclusion criteria, the inclusion criteria for the control group were as follows: not having a chronic spinal disorders and not having low back pain in the last week. Group II consisted of patients diagnosed with LSS and confirmed by MRI findings.

In addition to the general inclusion criteria, the inclusion criteria for the LSS group were as follows: having low back pain for more than 3 months and having low back pain intensity of 4 or more assessed with VAS.

There was not any additional inclussion criteria for Group III. The exclusion criteria of current study are; having any previous inner ear inflammation or vestibular disorders, having diabetes and being pregnant.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 50 years
* not having had lower extremity surgery
* not having a chronic spinal disorders
* not having low back pain in the last week
* having low back pain for more than 3 months
* having low back pain intensity of 4 or more assessed with VAS

Exclusion Criteria:

.having any previous inner ear inflammation or vestibular disorders .having diabetes and being pregnant.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group I consists of patient relatives and patients who applied to the outpatient clinic for another ailment.
  Group II consisted of patients diagnosed with LSS and confirmed by MRI findings.
  Participants who have undergone surgery due to LSS were included in Group III.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
reposition error | september 2020-february 2021
  Reposition error was asessed by measuring the difference in angles between the target position and the re-produced position. Target positions were 30º forward bending and 15º backward bending in sitting and standing positions. The target and the reproduced angles were measured with the iPhone tilt-meter application.
pain intensity | september 2020-february 2021
  . Pain intensity was assessed with the 10 cm horizontal Visual Analogue Scale (VAS) at target positions (during sitting and standing in combination with forward and backward bending)
flexibility of the TLF | september 2020-february 2021
  Flexibility of the TLF was evaluated with goniometric platform. The participant was asked to sit on a height-adjustable chair with the hip and knee flexed at 90º and the lumbar region in a neutral position. The goniometric platform was placed on the table in front of the participant. The therapist fixed the posterior superior iliac spines of the participant. And then participants were asked to hold the hands in front of the body (90° shoulder flexion) with a pen clamped between the hands. Participants were warned that the arms should follow the trunk rotation. Participants performed trunk rotation 3 times in the same direction and marked the point on the goniometric platform. The mean of the 3 measurements was calculated. The same protocol was repeated in the opposite direction.

CONTACTS AND LOCATIONS:
Overall Officials: Şule Şimşek, Phd, Principal Investigator — PhD faculty member
Locations (1):
- Denizli State Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AS, Cholewicki J, Reeves NP, Zazulak BT, Mysliwiec LW. Comparison of trunk proprioception between patients with low back pain and healthy controls. Arch Phys Med Rehabil. 2010 Sep;91(9):1327-31. doi: 10.1016/j.apmr.2010.06.004. PMID 20801248
- [Background] Sarioglu K, Pekyavas NO. A Comparison Between People With and Without Subacromial Impingement Syndrome and a New Method for Measuring Thoracolumbar Fascia Flexibility. J Chiropr Med. 2021 Mar;20(1):9-15. doi: 10.1016/j.jcm.2021.01.003. Epub 2021 May 12. PMID 34025300
- [Background] Noh KH, Oh JS, Yoo WG. Comparison of lumbar repositioning error according to different lumbar angles in a flexion pattern (FP) subgroup of patients with non-specific chronic low back pain. J Phys Ther Sci. 2015 Jan;27(1):293-4. doi: 10.1589/jpts.27.293. Epub 2015 Jan 9. PMID 25642094
- [Background] Georgy EE. Lumbar repositioning accuracy as a measure of proprioception in patients with back dysfunction and healthy controls. Asian Spine J. 2011 Dec;5(4):201-7. doi: 10.4184/asj.2011.5.4.201. Epub 2011 Nov 28. PMID 22164313